CLINICAL TRIAL: NCT01711034
Title: A Phase 1, Open-label, Multiple Dose Escalation Trial to Determine Safety and Tolerability of Once Daily OPB-111077 in Subjects With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 317-11-201
Record Dates: First submitted 2012-10-12; First posted 2012-10-22 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Solid Tumors
Keywords: Solid tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OPB-111077 (Experimental): In escalation stage of study, treatment with a once daily dose of OPB-111077 during cycles 1 and 2 on day 1, followed by 2-day treatment free interval, and then resuming daily dosing on day 4 through day 28. For cycle 3 and beyond, OPB-111077 will be administered for 28 continuous days per cycle until MTD is reached.
  In expansion portion of study, established dose of 250mg administered once daily for 28 consecutive days for each cycle. Patient in expansion are defined as those who meet eligibility criteria and have a diagnosed malignancy that is presumed to be susceptible to inhibition by OPB-111077
  Interventions: Drug: OPB-111077

INTERVENTIONS:
Drug: OPB-111077 — Dose escalation phase starting with dose of 100mg tablets on Day 1 and 4, and all remaining days of each 28 day cycle until disease progression or toxicity develops.
  Dose expansion phase starting with daily dosing of 250mg for 28 day consecutive day cycles.

SUMMARY:
The primary objective of this study is to determine the safe and tolerable dose level of OPB-111077 for patients with advanced cancer.

DETAILED DESCRIPTION:
The secondary objective of this study is to investigate the pharmacokinetic properties of OPB-111077; the pharmacodynamic effects of OPB-111077; the antitumor activity of OPB-111077 as assessed by RECIST or IMWG Uniform Response Criteria; and to explore whether PET responses correlate with other measures of clinical response.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically and/or cytologically confirmed advanced malignancy that is refractory to standard therapy or for which there are no standard treatment options available
* For oral or intravenous anticancer therapies, at least 4 weeks or 5 half-lives, whichever is shorter, need to have elapsed since the last dose
* Recovery from adverse effects of prior therapy at time of enrollment to

  o ≤ Grade 1 (excluding alopecia)
* Agreement to forego any other chemotherapy, immunotherapy, radiotherapy, or investigational drug while enrolled on this trial except hormonal therapy for prostate cancer or radiotherapy for symptomatic bone metastases known to be present at Screening
* Male or female subjects aged ≥ 18 years
* ECOG performance status ≤ 2
* Adequate organ function
* Life expectancy of ≥ 3 months following trial entry
* For women of childbearing potential, a negative serum pregnancy test result at Screening
* For women of childbearing potential or men whose sexual partners are women of childbearing potential, agreement to use 2 methods of adequate contraception prior to trial entry, for the duration of the trial, and for 90 days after the last dose of trial medication
* Signed and dated IRB-approved informed consent prior to any performance of protocol-specific screening procedures

Exclusion Criteria:

* Uncontrolled concurrent illness, including but not limited to: ongoing or active infection; uncontrolled heart, liver, kidney, or endocrine disorder
* Altered mental status, psychiatric illness, or social situation that would limit compliance with trial requirements and/or obscure trial results
* Immunocompromised state
* Known or evidence of chronic viral hepatitis (hepatitis B or C virus)
* Untreated or symptomatic brain metastasis, or subjects with leptomeningeal disease
* Inability to swallow oral meds or gastrointestinal disorder that might interfere with absorption of oral drugs
* Major surgery within 28 days of first receipt of trial drug
* Nursing or pregnant women
* ≥ Grade 1 neuropathy with pain or > Grade 2 neuropathy without pain (subjects with neuropathy caused by a previous regimen that is recovered to ≤ Grade 2 and stable without pain may be included)
* Food-effect sub-study (Part B) only: Pathologies or medical histories that might impair absorption and elimination.
* PET scan sub-study (Part C) only: Uncontrollable blood glucose or intolerance to PET scan procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2012-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of OPB-111077 | 28 Days
  AEs, Vital signs,Body weight, ECGs, Laboratory tests, Performance status

SECONDARY OUTCOMES:
To determine the pharmacokinetics of OPB-111077 | 28 Days
  The following PK parameters for Food-effect Sub-study (Cmax, AUCtau,AUCt, tmax, CLss/F and t1/2,z) will be determined using a non-compartmental approach for OPB-111077 and selected metabolites after single (Cycle 1, Day 1) and multiple daily doses (Cycle 2, Day 1).
Pharmacodynamic profile | 28 Days
  Study drug effects on STAT3 phosphorylation in response to IL-6 will be measured in PBMCs from subjects treated with OPB-111077.
Antitumor effects | Assessments will be conducted at Screening, Cycle 3, every 2 cycles (+/- 1 week) thereafter, at the Final/Early Termination Visit, and at the 30-day Follow-up Visit.
  Subjects with measurable disease will be assessed by RECIST Assessments will be conducted at Screening, Cycle 3, every 2 cycles (+/- 1 week) thereafter, at the Final/Early Termination Visit, and at the 30-day Follow-up Visit.
To determine the MTD of OPB-111077 | Within the first cycle [28 days].
  The highest dose at which fewer than 2 of 6 subjects experience DLT during the first 28 day cycle.
PET Sub-study (Part C) | 2 weeks
  A sub-study of up to 24 patients with PET-avid tumors where additional PET scans are performed to explore intra-subject PET activity.
Food-effect Sub-study (Part B) | 11 days
  An open-label, two-period crossover arm, for pre-selected study sites to determine the effect of food on the rate and extent of absorption (PK) following single dose 250mg OPB-111077.

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Rock, MD, PhD, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (1):
- San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tolcher A, Flaherty K, Shapiro GI, Berlin J, Witzig T, Habermann T, Bullock A, Rock E, Elekes A, Lin C, Kostic D, Ohi N, Rasco D, Papadopoulos KP, Patnaik A, Smith L, Cote GM. A First-in-Human Phase I Study of OPB-111077, a Small-Molecule STAT3 and Oxidative Phosphorylation Inhibitor, in Patients with Advanced Cancers. Oncologist. 2018 Jun;23(6):658-e72. doi: 10.1634/theoncologist.2017-0325. Epub 2018 Mar 6. PMID 29511132